CLINICAL TRIAL: NCT07027878
Title: JET Enhanced Thrombectomy Intervention Registry - JETi Registry
Brief Title: JETi Lower Extremity Venous Thrombosis
Acronym: JETiRegistry
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10433 Venous
Record Dates: First submitted 2025-06-05; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Venous Thrombosis
Keywords: ABT - CIP -10433; Venous Thrombosis; Thrombectomy intervention
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JETi™ Hydrodynamic Thrombectomy System: Subjects who were treated with JETi™ Hydrodynamic Thrombectomy System were included.
  Interventions: Device: JETi lower extremity venous thrombosis

INTERVENTIONS:
Device: JETi lower extremity venous thrombosis — The JETi System is a hydro-mechanical aspiration system, intended for the removal of intravascular thrombus. The system comprises of the JETi Catheter (6F or 8F), JETi Pump Set, JETi Saline Drive Unit (SDU), JETi Accessory Cart, JETi Suction tubing and JETi Non-Sterile Canister Set. The JETi System is designed to continuously aspirate thrombotic material into the catheter, where a high-pressure stream of saline within the catheter tip macerates the thrombus as it is aspirated.

SUMMARY:
The JETi Registry is a prospective, single-arm, multicenter study to collect real-world data on the safety, performance, and clinical benefits of the JETi System for the treatment of acute and subacute thrombosis in the peripheral vasculature. This is a post-market study that will register approximately 280 subjects at approximately 30 centers globally. Subjects participating in this registry will be followed through their 12-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was treated or is expected to be treated for acute/subacute thrombosis, as determined by the investigator, in the peripheral vasculature with the JETi Hydrodynamic Thrombectomy System.
2. Subject or legally authorized representative must provide written informed consent.
3. Subject must be ≥ 18 years of age.

Exclusion Criteria:

1. Subject has previously been registered in the JETi Registry in the last 12 months unless treated in the contralateral limb/different anatomy; patients treated in the contralateral limb/different anatomy within the last 12 months may re-enroll in the study.
2. Subject is currently participating in another drug or device clinical investigation.
3. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the past 20 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the patient population undergoing percutaneous treatment of thrombosis in the peripheral vascular system will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Composite of JETi-related major adverse events (MAEs) | Up to 30 days post-index procedure
  Composite of JETi-related MAEs up to 30 days post-JETi procedure, defined as the following JETi-related events adjudicated by a clinical event committee (CEC):
  1. death,
  2. symptomatic pulmonary embolism (PE),
  3. major bleeding
  4. re-thrombosis of JETi-treated vessel(s).
Percent of treated vessel(s) with ≥ 75% venous thrombus reduction via modified Marder score. The independent imaging core laboratory will be responsible for assessing this endpoint. | Perioperative/Periprocedural
  Percent of treated vessel(s) with ≥ 75% venous thrombus reduction via modified Marder from pre-JETi venogram to final venogram (post-JETi AND after any/all adjunctive therapies to treat underlying culprit lesions)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (21):
  - HonorHealth, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - PIH Good Samaritan, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University Hospital and Clinics, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - ClinRé, Thornton, Colorado
  - St. Mary Medical Center, Hobart, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Louisville, Louisville, Kentucky
  - Southoast Hospital, Fall River, Massachusetts
  - Henry Ford Detroit, Detroit, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Hendrick Medical Center, Abilene, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Charleston Area Medical Center, Charleston, West Virginia
- Royal Perth Hospital, Perth, Australia
- Hôpital Saint-François d'Assise, Québec, Quebec, Canada
- Germany (7):
  - University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Marien Hospital Herne, Herne, North Rhine-Westphalia
  - Klinikum Hochsauerland, Arnsberg
  - Evangelisches Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Sankt Gertrauden Krankenhaus, Berlin
  - Medizinische Einrichtungen der Universität zu Köln, Cologne
  - Universitätsklinikum Giessen, Giessen

DOCUMENTS (1):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT07027878/Prot_000.pdf